CLINICAL TRIAL: NCT04950426
Title: Impact of Post-Traumatic Stress Disorder Treatment by Reconsolidation Therapy on Fibromyalgia Syndrome
Acronym: PTSD-FMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000312-36
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia Syndrome; Posttraumatic Stress Disorder
MeSH Terms: conditions — Fibromyalgia; Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with reconsolidation therapy (Experimental): Patient will take propranolol once a week during 6 weeks. The dosage of propranolol: 1 mg/kg propranolol form: tablet
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — One administration of propranolol, once a week during six weeks. Reading by the participant of his/her traumatic story, 75 minutes (+/- 15 min) after propranolol intake.

SUMMARY:
The aim of the study is to demonstrate a significant improvement in quality of life specific to patients with fibromyalgia syndrome in patients with fibromyalgia syndrome with comorbid posttraumatic stress disorder, treated with reconsolidation blockade.

Patients receive a treatment with propranolol associated with reconsolidation blockade of traumatic story once a week during 6 weeks, with evaluation at inclusion and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old
* Diagnosis of fibromyalgia syndrome according to ACR 2016 criteria
* PCL-5 > 44 suggesting the presence of a comorbid post-traumatic stress disorder
* Meet the DSM-5 criteria for post-traumatic stress disorder secondary to exposure to a traumatic event according to DSM-5 criteria, both unique or repeated and regardless of the date or location of the traumatic event.
* Pain relief treatment and/or psychotropic treatment stabilized for a period greater than or equal to two months.
* Signature of a consent form
* Patient able to understand and read french

Exclusion Criteria:

* Psychotic disorders
* Unstable bipolar disorder
* Patients with a systolic blood pressure < 100 mmHg or heart rate < 55 as established during the initial visit
* Significant anormal ECG
* Medical contraindication to taking propranolol
* Adverse reactions or previous intolerances to a beta blocker
* Current intake of another beta blocker which can not be stopped during the protocol, regardeless the galenic.
* Current intake of a drug with potential contraindication with the propranolol, according to the summary of product characteristics of the propranolol.
* Patient under legal protection, under guardianship or under curatorship
* Patient having suffered a head trauma for less than a year or with clinical symptoms and neurological sequelae
* Known severe suicide risk (MINI-S and medical exam)
* Current opioid addiction or alcohol dependence
* Patients treated for less than 2 months with antidepressants or painkillers
* Patients unafiliated to a social health care
* Woman who is pregnant or breast-feeding or whithout efficient contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Significant improvement in quality of life specific to patients with fibromyalgia syndrome in patients with fibromyalgia syndrome with comorbid posttraumatic stress disorder, treated with reconsolidation therapy. | 3 months
  Modification in quality of life in patients with fibromyalgia syndrome measured by the Fibromyalgia Impact Measurement Questionnaire (FIQ).
  FIQ minimal value:0 (minimum impact) FIQ maximal value: 100 (maximal impact)

CONTACTS AND LOCATIONS:
Overall Officials: Nematollah Jaafari, Professor, Principal Investigator — Centre Hospitalier Henri Laborit
Locations (2):
- France (2):
  - Centre Hospitalier Henri Laborit, Poitiers
  - Centre Hospitalier Nord-Deux-Sèvres, Thouars

IPD SHARING:
Plan to Share IPD: No